CLINICAL TRIAL: NCT04689815
Title: Measurable-residual Disease (MRD) Monitoring of Nucleophosmin 1 (NPM1)-Mutated Acute Myeloid Leukaemia (AML) and Pre-emptive Therapy With Oral Arsenic Trioxide-based Regimen
Brief Title: Oral Arsenic Trioxide for NPM1-mutated AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPM1001
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: NPMc+ AML
Keywords: NPM1 mutation; Acute myeloid leukemia; Oral arsenic trioxide
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral arsenic trioxide-Azacitidine (Experimental): 12 monthly cycles of oral arsenic trioxide (oral-As2O3) (Arsenol ®) (5-10mg per day, from days 1-7 per cycle), ascorbic acid (1g per day, from days 1 - 7 per cycle) plus azacitidine (75mg/m2 per day subcutaneously, from days 1 to 3 per cycle).
  Interventions: Drug: Oral Arsenic Trioxide Formulation

INTERVENTIONS:
Drug: Oral Arsenic Trioxide Formulation — Eligible subjects with NPM1 MRD positivity will receive oral arsenic trioxide (oral-As2O3) (Arsenol ®) (5-10mg per day, from days 1-7 per cycle), ascorbic acid (1g per day, from days 1 - 7 per cycle) plus azacitidine (75mg/m2 per day subcutaneously, from days 1 to 3 per cycle). Each cycle of oral-As2O3 plus azacitidine will be given once every 28 days. The total duration of treatment is 12 months (12 cycles). Treatment will be day-care and outpatient based. Reduction in the dosage and duration of oral-As2O3 is required if the subject is experiencing adverse events (AEs). In case of grade 3 or above toxicity, the dosage of oral-As2O3 will be reduced to 5mg per day.
  Other Names: Arsenol

SUMMARY:
A prospective open-label phase 2 study will be designed to assess the efficacy of oral arsenic trioxide plus azacitidine in preventing relapses in patients with NPM1-mutant AML. After screening and eligibility assessment, patients will receive treatment with oral arsenic trioxide plus azacitidine for 12 months. The recruitment period will last for 24 months and it will take approximately 36 months for study completion.

DETAILED DESCRIPTION:
Eligible subjects with NPM1 MRD positivity will receive oral arsenic trioxide (oral-As2O3) (Arsenol ®) (5-10mg per day, from days 1-7 per cycle), ascorbic acid (1g per day, from days 1 - 7 per cycle) plus azacitidine (75mg/m2 per day subcutaneously, from days 1 to 3 per cycle). Each cycle of oral-As2O3 plus azacitidine will be given once every 28 days. The total duration of treatment is 12 months (12 cycles). Treatment will be day-care and outpatient based. Reduction in the dosage and duration of oral-As2O3 is required if the subject is experiencing adverse events (AEs). In case of grade 3 or above toxicity, the dosage of oral-As2O3 will be reduced to 5mg per day. Changes or interruption in dosages, their dates and time points will be recorded on the dosage administration record and the electronic case report form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years
2. Diagnosis of AML with NPM1 mutation
3. Positive MRD for NPM1 mutation after completion of consolidation in transplant-ineligible patients
4. Positive MRD for NPM1 mutation after allogeneic HSCT
5. bilirubin ≤ 1.5 x upper limit normal (ULN); alanine aminotransferase (ALT) ≤ 2 x ULN or aspartate aminotransferase (AST) ≤ 2 x ULN; and prothrombin time versus control <3 seconds at screening
6. Glomerular filtration rate ≥ 50 mL/min (by MDRD equation or Cockcroft-Gault formula)
7. Corrected QT interval (QTc) (by Framingham formula) <500ms.
8. Able to give a written informed consent and fully comply to the requirements of the study.

Exclusion Criteria:

1. Patients on other investigational therapies
2. Prior exposure to azacitidine, decitabine or arsenic trioxide
3. Uncontrolled graft-versus-host disease (GVHD)
4. Eastern Cooperative Oncology Group (ECOG) performance status > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of NPM1 MRD negativity. | 36 months
  This is defined as undetectable NPM1 mutant transcript with RQ-PCR on both the PB and BM following treatment, at a limit of detection of 10^-5.

SECONDARY OUTCOMES:
Duration of response | 36 months
  defined as the time from achievement of undetectable NPM1 MRD to Documented molecular recurrence (defined as detectable MRD on PB or BM at a limit of detection of 10^5.
Leukaemia-free survival (LFS) | 36 months
  This is defined as the time, in months, from the start of oral-As2O3 plus azacitidine to morphologic relapse of AML.
Safety of oral-As2O3 plus azacitidine, assessed using the common toxicity criteria for adverse events (CTCAE) version 5.0. | 36 months
  The incidence of treatment emergent adverse events will be determined as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Gill, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papaemmanuil E, Gerstung M, Bullinger L, Gaidzik VI, Paschka P, Roberts ND, Potter NE, Heuser M, Thol F, Bolli N, Gundem G, Van Loo P, Martincorena I, Ganly P, Mudie L, McLaren S, O'Meara S, Raine K, Jones DR, Teague JW, Butler AP, Greaves MF, Ganser A, Dohner K, Schlenk RF, Dohner H, Campbell PJ. Genomic Classification and Prognosis in Acute Myeloid Leukemia. N Engl J Med. 2016 Jun 9;374(23):2209-2221. doi: 10.1056/NEJMoa1516192. PMID 27276561
- [Background] Patel JP, Gonen M, Figueroa ME, Fernandez H, Sun Z, Racevskis J, Van Vlierberghe P, Dolgalev I, Thomas S, Aminova O, Huberman K, Cheng J, Viale A, Socci ND, Heguy A, Cherry A, Vance G, Higgins RR, Ketterling RP, Gallagher RE, Litzow M, van den Brink MR, Lazarus HM, Rowe JM, Luger S, Ferrando A, Paietta E, Tallman MS, Melnick A, Abdel-Wahab O, Levine RL. Prognostic relevance of integrated genetic profiling in acute myeloid leukemia. N Engl J Med. 2012 Mar 22;366(12):1079-89. doi: 10.1056/NEJMoa1112304. Epub 2012 Mar 14. PMID 22417203
- [Background] Ivey A, Hills RK, Simpson MA, Jovanovic JV, Gilkes A, Grech A, Patel Y, Bhudia N, Farah H, Mason J, Wall K, Akiki S, Griffiths M, Solomon E, McCaughan F, Linch DC, Gale RE, Vyas P, Freeman SD, Russell N, Burnett AK, Grimwade D; UK National Cancer Research Institute AML Working Group. Assessment of Minimal Residual Disease in Standard-Risk AML. N Engl J Med. 2016 Feb 4;374(5):422-33. doi: 10.1056/NEJMoa1507471. Epub 2016 Jan 20. PMID 26789727
- [Background] Balsat M, Renneville A, Thomas X, de Botton S, Caillot D, Marceau A, Lemasle E, Marolleau JP, Nibourel O, Berthon C, Raffoux E, Pigneux A, Rodriguez C, Vey N, Cayuela JM, Hayette S, Braun T, Coude MM, Terre C, Celli-Lebras K, Dombret H, Preudhomme C, Boissel N. Postinduction Minimal Residual Disease Predicts Outcome and Benefit From Allogeneic Stem Cell Transplantation in Acute Myeloid Leukemia With NPM1 Mutation: A Study by the Acute Leukemia French Association Group. J Clin Oncol. 2017 Jan 10;35(2):185-193. doi: 10.1200/JCO.2016.67.1875. Epub 2016 Nov 14. PMID 28056203
- [Background] Dillon R, Hills R, Freeman S, Potter N, Jovanovic J, Ivey A, Kanda AS, Runglall M, Foot N, Valganon M, Khwaja A, Cavenagh J, Smith M, Ommen HB, Overgaard UM, Dennis M, Knapper S, Kaur H, Taussig D, Mehta P, Raj K, Novitzky-Basso I, Nikolousis E, Danby R, Krishnamurthy P, Hill K, Finnegan D, Alimam S, Hurst E, Johnson P, Khan A, Salim R, Craddock C, Spearing R, Gilkes A, Gale R, Burnett A, Russell NH, Grimwade D. Molecular MRD status and outcome after transplantation in NPM1-mutated AML. Blood. 2020 Feb 27;135(9):680-688. doi: 10.1182/blood.2019002959. PMID 31932839
- [Background] Martelli MP, Gionfriddo I, Mezzasoma F, Milano F, Pierangeli S, Mulas F, Pacini R, Tabarrini A, Pettirossi V, Rossi R, Vetro C, Brunetti L, Sportoletti P, Tiacci E, Di Raimondo F, Falini B. Arsenic trioxide and all-trans retinoic acid target NPM1 mutant oncoprotein levels and induce apoptosis in NPM1-mutated AML cells. Blood. 2015 May 28;125(22):3455-65. doi: 10.1182/blood-2014-11-611459. Epub 2015 Mar 20. PMID 25795919
- [Background] El Hajj H, Dassouki Z, Berthier C, Raffoux E, Ades L, Legrand O, Hleihel R, Sahin U, Tawil N, Salameh A, Zibara K, Darwiche N, Mohty M, Dombret H, Fenaux P, de The H, Bazarbachi A. Retinoic acid and arsenic trioxide trigger degradation of mutated NPM1, resulting in apoptosis of AML cells. Blood. 2015 May 28;125(22):3447-54. doi: 10.1182/blood-2014-11-612416. Epub 2015 Mar 23. PMID 25800051
- [Background] Chau D, Ng K, Chan TS, Cheng YY, Fong B, Tam S, Kwong YL, Tse E. Azacytidine sensitizes acute myeloid leukemia cells to arsenic trioxide by up-regulating the arsenic transporter aquaglyceroporin 9. J Hematol Oncol. 2015 May 8;8:46. doi: 10.1186/s13045-015-0143-3. PMID 25953102